CLINICAL TRIAL: NCT06881914
Title: Enhancing Life Quality in Community-dwelling Older Omanis by Telling Their Life Story and Creating Life-story Book
Brief Title: Enhancing Life Quality in Community-Dwelling Older Omanis by Telling Their Life Story
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sultan Qaboos University (Other)
Responsible Party: Principal Investigator, Moon Fai Chan, PhD, Associate Professor, Sultan Qaboos University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MREC#2028
Record Dates: First submitted 2025-03-07; First posted 2025-03-18 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Healthy Older Adults
Keywords: Depression; Life satifaction; Quality of life; Older adults
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: Intervention group: There were 5 sessions for the intervention group. All sessions took place in the participant's home. In the first 4 sessions, the participant was asked to share their childhood, adolescence, adulthood, and current stage. Transcripts were prepared and compiled following the completion of the interviews. Before printing, participants were asked to add their selected pictures to the life-story book. In the 5th session, they received their life story-story books. A self-report questionnaire was used in every session to collect participants' quality of life, life satisfaction, and depression scores.
  Control group: The control group had 5 sessions, and participants' quality of life, life satisfaction, and depression scores were collected at each interview only.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (No Intervention): Five sessions took place at the participants' homes. A self-report questionnaire was used in every session to collect participants' quality of life, life satisfaction, and depression scores.
- Life-story review (Experimental): The life-story review intervention consisted of five sessions, during which participants shared their life experiences/stories and compiled them into a life-story book. In each session, a self-report questionnaire was administered to assess participants' quality of life, life satisfaction, and levels of depression.
  Interventions: Behavioral: Intervention group:

INTERVENTIONS:
Behavioral: Intervention group: — There were 5 sessions for the intervention group. All sessions took place in the participant's home. The first 4th sessions involved participant sharing a particular time of their life event, such as childhood, adolescence, adulthood, and the current stage. Transcripts were prepared and compiled following the completion of the interviews. The participants will proofread their life-story book before sending it for printing. In the 5th session, they were given their life storybooks. A self-report questionnaire was used in every session to collect participants' quality of life, life satisfaction, and depression scores.
  Arms: Life-story review

SUMMARY:
This study investigates whether sharing life stories and creating life-story books can enhance the quality of life and life satisfaction and reduce depression in older adults. The primary research question is:

Did the quality of life, life satisfaction, and levels of depression improve more for participants in the intervention group compared to those in the control group?

Participants will be divided into two groups:

* Intervention group: These participants will share life stories and create life-story books.
* Control group: These participants will not share life stories or create life-story books.

DETAILED DESCRIPTION:
Background: The main goal of this study is to investigate whether telling their life stories and developing a life-story book intervention affects a group of Omani older adults' quality of life, life satisfaction, and depression symptoms.

Methods: In Oman, a randomized controlled trial with repeated measures was conducted to evaluate the impact of the intervention. 75 older individuals were randomly assigned to either the intervention group (n = 38) or the control group (n = 37). Baseline demographic data were collected as an initial reference point. To comprehensively assess changes over time, participants' depression levels, life satisfaction, and overall quality of life were measured at multiple time points: weeks 1, 2, 3, 4, and 8. This longitudinal design allowed for a nuanced analysis of intervention effects across different implementation phases.

This study believes that participants in the 8-week trial of the life-story review intervention were successful in reducing depression and improving life satisfaction and quality of life in the older population. Healthcare professionals can use such interventions to enhance older persons' mental health and well-being.

ELIGIBILITY:
Inclusion Criteria:

* aged 60-90;
* depressive symptoms score between 5 and 10;
* able to sign the consent form;
* able to speak Arabic or English;
* able to communicate without the need for a hearing aid.

Exclusion Criteria:

* using hypnotics, sedatives, antidepressants, anticholinergics, antihistamines, tranquilizers, or melatonin for sleep;
* having a medical diagnosis of Parkinson's, dementia, Alzheimer's disease, or a serious mental problem;
* Participants assigned to the intervention group who did not want to be audio recorded.

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the depression scores (GDS-15) at 8 weeks | From enrollment to the end of intervention at 8 weeks.
  The Geriatric Depression Scale (GDS-15), Arabic version, was used to collect depression scores. It comprises 15 closed-ended questions regarding how the elderly participants felt during the previous week. Zero indicates no depressive symptoms, and 15 indicates severe depressive symptoms.

SECONDARY OUTCOMES:
Change from baseline in the life satisfaction score at 8 weeks | From enrollment to the end of treatment at 8 weeks
  The Arabic version of the Satisfaction with Life Scale (SWLS) was used to collect older adults' degrees of life satisfaction. The SWLS consists of 5 items with response options ranging from 1 (strongly disagree) to 7 (strongly agree), and it has good reliability (a = 0.86). A total score of 35 indicates greater life satisfaction; a score of 5 indicates poor life satisfaction.
Change from baseline in the quality of life score at 8 weeks | From enrollment to the end of treatment at 8 weeks.
  World Health Organization Quality of Life Questionnaire (WHOQoL-BREF) The World Health Organization Quality of life questionnaire, The WHOQoL-BREF, in Arabic, assesses older persons' health-related quality of life. It is a 26-item test with a 5-point Likert-type scale; a higher score would suggest a higher quality of life regarding the environment, social interactions, psychology, and physical health.

CONTACTS AND LOCATIONS:
Overall Officials: Moon Fai Chan, PhD, Principal Investigator — Sultan Qaboos University, Department of Family Medicine and Public Health, Muscat, Oman
Locations (1):
- Sultan Qaboos University Hospital, Muscat, Muḩāfaz̧at Masqaţ, Oman

IPD SHARING:
Plan to Share IPD: No
Each participant's life story sharing information is private and confidential, so they did not allow sharing this information with other parties.